CLINICAL TRIAL: NCT00811564
Title: An Evaluation of the Fixed Combination Brimonidine Tartrate 0.2%/ Timolol Maleate 0.5% to Latanoprost 0.005% in Glaucoma or Ocular Hypertension Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Medical Affairs Director, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMA-COM-08-008
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-08

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Timolol; Ophthalmic Solutions; Brimonidine Tartrate, Timolol Maleate Drug Combination; Latanoprost

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Active Comparator): Fixed combination of brimonidine tartrate 0.2%/timolol maleate 0.5% ophthalmic solution
  Interventions: Drug: fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% ophthalmic solution
- 2 (Active Comparator): Latanoprost 0.005% ophthalmic solution
  Interventions: Drug: latanoprost 0.005%

INTERVENTIONS:
Drug: fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% ophthalmic solution — 1 drop of study medication taken approximately 12 hours apart, dosed 2 times a day
  Other Names: Combigan™
  Arms: 1
Drug: latanoprost 0.005% — 1 drop of study medication taken once daily
  Other Names: Xalatan™
  Arms: 2

SUMMARY:
A three-month evaluation comparing the safety and efficacy of a fixed combination of 0.2% brimonidine tartrate/0.5% timolol maleate with that of latanoprost 0.005%, a prostaglandin analogue in glaucoma or ocular hypertension subjects

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age;
2. Give written informed consent;
3. Be in good general health as determined by your doctor;
4. Have a diagnosis of unilateral or bilateral glaucoma or ocular hypertension;
5. If you are a female of child bearing potential, you must be willing to practice effective contraception for the duration of the study (i.e., abstinence, spermicide, condoms, or birth control pills);
6. Understand the study instructions, and be able to follow the study instructions; and
7. Be likely to complete the entire study period (12 weeks), including all regularly scheduled study visits.

Exclusion Criteria:

1. Have any active ocular disease other than glaucoma or ocular hypertension that would interfere with study interpretation;
2. Any systemic disease or clinical evidence of any condition which would make the subject, in the opinion of the investigator, unsuitable for the study or could potentially confound the study results; and
3. Concurrent participation or prior participation in any investigational drug or device study within the last 30 days prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Slingerlands, New York, United States

REFERENCES:
- [Derived] Katz LJ, Rauchman SH, Cottingham AJ Jr, Simmons ST, Williams JM, Schiffman RM, Hollander DA. Fixed-combination brimonidine-timolol versus latanoprost in glaucoma and ocular hypertension: a 12-week, randomized, comparison study. Curr Med Res Opin. 2012 May;28(5):781-8. doi: 10.1185/03007995.2012.681036. Epub 2012 Apr 25. PMID 22458918

RESULTS

PARTICIPANT FLOW:
Groups:
- Fixed Combination of Brimonidine Tartrate 0.2%/Timolol Maleate: Fixed combination of brimonidine tartrate 0.2%/timolol maleate 0.5% ophthalmic solution
- Latanoprost 0.005% Ophthalmic Solution: Latanoprost 0.005% ophthalmic solution
Period: Overall Study
Arm/Group | Fixed Combination of Brimonidine Tartrate 0.2%/Timolol Maleate | Latanoprost 0.005% Ophthalmic Solution
Started | 73 | 75
Completed | 64 | 73
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Combination of Brimonidine Tartrate 0.2%/Timolol Maleate | Latanoprost 0.005% Ophthalmic Solution | Total
Number analyzed (Participants) | 73 | 75 | 148
Age Continuous [Median (Full Range); unit: years] | 65 [27 to 88] | 65 [33 to 87] | 65 [27 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 86
  Male | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at Week 12
Description: Mean IOP at week 12. IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Week 12
Population: Intent-to-treat, which included all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mm Hg)
Arm/Group | Fixed Combination of Brimonidine Tartrate 0.2%/Timolol Maleate | Latanoprost 0.005% Ophthalmic Solution
Number analyzed (Participants) | 73 | 75
Millimeters of mercury (mm Hg) | 17.75 (2.878) | 17.90 (3.943)

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized AND treated.
Arm/Group | Fixed Combination of Brimonidine Tartrate 0.2%/Timolol Maleate | Latanoprost 0.005% Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/73 | 1/75
Other Adverse Events (participants affected / at risk) | 8/73 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Combination of Brimonidine Tartrate 0.2%/Timolol Maleate (N=73) | Latanoprost 0.005% Ophthalmic Solution (N=75)
Anemia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Combination of Brimonidine Tartrate 0.2%/Timolol Maleate (N=73) | Latanoprost 0.005% Ophthalmic Solution (N=75)
Eye irritation (Eye disorders) | 4 | 0
Pain eye (Eye disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo